CLINICAL TRIAL: NCT03118622
Title: A Comparison of Pentax AWS Videolaryngoscopy and Macintosh Laryngoscopy for Orotracheal Intubation in Children: a Randomized Controlled Trial
Brief Title: Pentax Videolaryngoscopy in Children
Acronym: Pentax
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, Clinical assistant professor, Ajou University School of Medicine
Other Study IDs: AJIRB-TEMP-TEMP-17-170
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Intubation;Difficult

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pentax group: Intubation using Pentax
  Interventions: Device: Pentax
- Macintosh group: Intubation using Macintosh

INTERVENTIONS:
Device: Pentax — Intubation using Pentax video laryngoscope in Pentax group
  Groups: Pentax group

SUMMARY:
Comparison of Intubation using Pentax (Pentas AWS, Pentax, Tokyo, Japan) and Macintoch in pediatric patients

DETAILED DESCRIPTION:
Pentax video laryngoscope (Pentas AWS, Pentax, Tokyo, Japan) is one of indirect optical laryngoscopes which is recently developed. Several studies have shown that the Pentax-AWS® provides full views of the glottis in the majority of patients. It makes successful tracheal intubation in patients after failed intubation using a Macintosh laryngoscope.

In pediatric patients who is expected to be difficult to intubate, Pentax makes successful intubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1, 2
* Scheduled surgery under general anesthesia

Exclusion Criteria:

* Intraoral disease
* Congenital anomaly
* C-spine injury
* Patients who need Rapid sequence induction

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Intubation time | less than 10 minute
  from laryngoscope pass incisors to end tidal CO2 appears

SECONDARY OUTCOMES:
Intubation difficulty score | less than 10 minute
  IDS parameter is Number of attempts > 1 = N1 Number of operators >1 = N2 Number of alternative techniques = N3 Cormack and Lehane grade minus 1 = N4 Operator perception of lifting force required Normal N5 = 0 Greater than in routine practice N5=1 Laryngeal pressure applied Not applied N6=0 Applied N6=1 Vocal core mobility Abduction N7=0 Adduction &/or impending tube passage N7=1 Total IDS = sum of scores N1~N7

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yi IK, Kwak HJ, Kim KM, Ahn SH, Lee SY, Kim JY. Comparison of Pentax Airway Scope and Macintosh laryngoscope for orotracheal intubation in children: A randomised non-inferiority trial. Acta Anaesthesiol Scand. 2019 Aug;63(7):853-858. doi: 10.1111/aas.13368. Epub 2019 Mar 22. PMID 30900242